CLINICAL TRIAL: NCT01635205
Title: Efficacy of Paraspinous Anesthetic Block in Patients With Chronic Pelvic Pain Non-Responsive to Pharmacological Treatment
Brief Title: Paraspinous Anesthetic Block for Non-Responsive Pelvic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GPPG 110082
Record Dates: First submitted 2011-12-17; First posted 2012-07-09 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Paraspinous Block; Pelvis Pain Chronic
Keywords: Paraspinous block; Non-responsive chronic pelvic pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paraspinous block (Experimental): Paraspinous anesthetic block in the thoracolumbar region, in sensitized segments
  Interventions: Procedure: paraspinous anesthetic block
- control (Sham Comparator): Subcutaneous puncture with no anesthetic effect
  Interventions: Procedure: subcutaneous puncture with no anesthetic effect

INTERVENTIONS:
Procedure: paraspinous anesthetic block — Paraspinous anesthetic block with lidocaine 1% in sensitized segments of the thoracolumbar region
  Arms: paraspinous block
Procedure: subcutaneous puncture with no anesthetic effect — Subcutaneous puncture with injection needle (no substance will be injected)
  Arms: control

SUMMARY:
This study examines randomized triple-blind clinical trial and the efficacy of paraspinous anesthetic block on the treatment of chronic pelvic pain in patients non-responsive to pharmacological management. Sixty patients will be randomly divided and allocated into group intervention (paraspinous anesthetic block) and control (placebo procedure in subcutaneous tissue).

DETAILED DESCRIPTION:
Patients will be allocated into one of two groups (intervention or placebo), and will be submitted to the corresponding procedure (paraspinous anesthetic block or placebo puncture in subcutaneous tissue). In the first appointment, pain will be measured with the VAS (Visual Analogue Scale); quality of life and function basal level will be evaluated by scales SF-36 (Medical Outcome Short-Form (36)Health Survey)and FSFI (Female Sexual Function Index), in Portuguese validated versions. Procedure will be realized as planned for each group.

Second appointment will occur one week after the procedure, and VAS scale will be applied.

Third appointment will occur in one month. VAS scale will be applied again,and procedure will be repeated if patient does not have a reduction of at least 30% of pain.

Next consultations will occur at two months, three months, four months and five months, with application of VAS scale to keep monitoring evolution of pain.

At six months of study, VAS scale will be applied along with SF-36 and FSFI questionnaires, to evaluate improvement in pain and in quality of life and function level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign pelvic pain non-responsive to pharmacological treatment, lasting at least 6 months, located in the anatomic pelvis, anterior abdominal wall, infra-umbilical region, lumbossacral region or buttocks. Pain must be hard enough to cause functional impairment or to motivate medical counseling. The absence of physical findings does not decreases the importance of pain, nether excludes the possibility of pelvic pathology.

Exclusion Criteria:

* Patients who do not want to take part in the study
* Age under 18 years old
* Pelvic pain lasting less than 6 months
* Relief or resolution of pain with pharmacological treatment
* Pain of neoplastic origin
* Known allergy or report of adverse reaction related to lidocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change of pain from baseline | Change of pain from baseline at one week, at one month, at two months, at three months, at four months, at five months and at six months
  Primary outcome is the reduction of pain, measured with the Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Improvement of scores in SF-36 scale | At baseline and at six months
  Quality of life will be evaluated with SF-36 scale at baseline and at six months, and scores will be compared at the end of the study.
Improvement of scores in the FSFI scale | At baseline and at six months
  Sexual function as a measure of functionality will be evalueted with the FSFI scale at baseline and at six months, and scores will be compared at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Rosa, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Antonio C Santos, doctor, Study Chair — Hospital de Clínicas de Porto Alegre; Ricardo F Savaris, doctor, Study Chair — Hospital de Clínicas de Porto Alegre; Vinícius A Amantéa, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] da Rosa KF, Amantea VA, dos Santos AC, Savaris RF. Efficacy of paraspinal anesthetic block in patients with chronic pelvic pain refractory to drug therapy: a randomized clinical trial. Rev Bras Ginecol Obstet. 2015 Mar;37(3):105-9. doi: 10.1590/SO100-720320150005201. PMID 25830642